CLINICAL TRIAL: NCT02883803
Title: Effects of Mesenchymal Stem Cells Administration on Organ Failure During Septic Shock: Phase II Randomized Comparator-controlled Study
Brief Title: Treatment of Severe Infections With Mesenchymal Stem Cells
Acronym: CHOCMSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRCI 2012/CHOCMSC-GIBOT/SKJ
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC (Experimental): Patients hospitalized in recovery unit and having a very severe septic shock with community origin (≥ 2 organ failures other than hemodynamic) since less than 12 hours, will receive 10^6/kg heterologous mesenchymal stem cells in 250 ml albumin 4%, infused for 30 minutes in central venous line.
  Interventions: Biological: Injection of mesenchymal stem cells
- Placebo (Sham Comparator): Patients hospitalized in recovery unit and having a very severe septic shock with community origin (≥ 2 organ failures other than hemodynamic) since less than 12 hours, will receive 250 ml albumin 4%, infused for 30 minutes in central venous line.
  Interventions: Biological: Injection of albumin alone

INTERVENTIONS:
Biological: Injection of mesenchymal stem cells — Injection of mesenchymal stem cells
  Arms: MSC
Biological: Injection of albumin alone — Injection of albumin alone
  Arms: Placebo

SUMMARY:
The main purpose at the early phase of septic shock on the evolution of organ failure judged by the SOFA (Sepsis Organ Failure Assessment score) score on Day 7 (or the day of death or the day of discharge from the intensive care unit if before Day 7) compared to SOFA score observed in patients in the control group. The secondary purpose is to assess the role of heterologous mesenchymal stem cells on the occurrence and duration of failure of each organ and on the mortality at day 28 and day 90. The safety of administration will be also assessed.

DETAILED DESCRIPTION:
Patients hospitalized in recovery unit and having a very severe septic shock with community origin (≥ 2 organ failures other than hemodynamic) since less than 12 hours, will receive 10^6/kg heterologous mesenchymal stem cells in 250 ml albumin 4%, infused for 30 minutes in central venous line or 250 ml albumin 4% alone.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock of community origin since less than 12 hours. The onset time of septic shock is the time of catecholamine introduction( adrenaline, noradrenaline, or dopamine > 8μg/kg/min)
* At least 2 organ failure other than hemodynamic
* Occurrence between Monday 8am and Friday 8am (for availability reasons of staff)
* Signature of informed consent (patient/close relative or reliable person)
* Affiliation to social security plan

Exclusion Criteria:

* Non-septic shock
* Nosocomial septic shock
* PaO2/FiO2 <100
* Pregnant or breast-feeding woman
* Brain death
* Dying person
* Therapeutic limitations
* Participation to another current interventional clinical trial or since less than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
SOFA score | Day 7 (or death day or day of recovery unit exit if before day 7)
  To assess the efficacy of a recovery treatment

SECONDARY OUTCOMES:
Number of living days without catecholamines | Day 28
Number of living days without mechanical ventilation | Day 28
Number of living days without dialysis | Day 28
Duration of residence time in recovery unit | Day of exit from recovery unit, up to 90 days
Mortality, across all causes | Day 28
Mortality, across all causes | Day 90
Administration safety (i.e. side effects) | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GIBOT, Principal Investigator — Service de Réanimation Médicale, Hôpital Central, 54035, Nancy Cedex
Locations (4):
- France (4):
  - Service de Réanimation Médicale, Hôpital Bocage, Dijon
  - Service de Réanimation Médicale, Hôpital Central, Nancy
  - Hôpital Hautepierre, Service de réanimation médicale, Strasbourg
  - UTCT, Hôpital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No